CLINICAL TRIAL: NCT04766749
Title: Remote Ischemic Preconditioning on the Prognosis of Patients With Elective PCI Using Drug-coated Balloon
Acronym: RIPC-DCB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HenanICE202104
Record Dates: First submitted 2021-02-10; First posted 2021-02-23 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Before the operation, the nurse chooses the patient to perform RIPC or not according to a predefined random method, and then the operation is performed by the operator.
  The operator did not know if the patient had undergone RIPC. Outcome evaluators also did not know the grouping of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 40 minutes before PCI by the nurse to the patient RIPC operation (RIPC is delivered with a standard blood pressure cuff placed on the upper thigh. The cuffs are inflated to 200 mm Hg and keep inflated for 5 minutes,Then deflated to 0 mmHg and keep uninflated for 5 minutes, This cycle is repeated four times), and then do regular PCI operation
  Interventions: Other: RIPC
- Control (No Intervention): A standard cuff is placed on the patient's thigh by the nurse 40 minutes before PCI but it is not inflated. PCI is performed 40 minutes later

INTERVENTIONS:
Other: RIPC — RIPC is delivered with a standard blood pressure cuff placed on the upper thigh. The cuffs are inflated to 200 mm Hg and keep inflated for 5 minutes,Then deflated to 0 mmHg and keep uninflated for 5 minutes, This cycle is repeated four times
  Arms: Experimental

SUMMARY:
Drug-coated balloon is being used more and more widely for the advantage of intervention without implantation.

But the balloon needs to be released long enough to be effective. Prolonged balloon dilation resulting in the cessation of blood flow in the distal vessels, especially large vessels, may result in severe ischemia in the patient.

RIPC can enhance patients' tolerance to ischemic events, so we believe that RIPC application before the use of drug balloon for PCI can improve patients' ischemic symptoms, thus increasing the release time of drug balloon and improving the effect.

DETAILED DESCRIPTION:
Some patients receiving PCI cannot tolerate the symptoms of myocardial ischemia caused by the release of the drug balloon for a long time and even lead to the occurrence of adverse events.RIPC was found to improve tolerance to myocardial ischemia in patients.

At the same time, it can open collateral circulation and improve the tolerance of myocardial ischemia in patients.Therefore, this study designed a parallel control group. The experimental group was treated with RIPC before PCI, while the control group was not treated before PCI.

The operator does not know whether the patient has undergone RIPC or not, and the operator decides the time of drug balloon release according to the symptoms of the patient during the operation.Angiography was performed at 6 months, and QCA was used to determine late lumen loss at 1 year.The 1-year incidence of target lesion failure events was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diameter stenosis>=50% by visual estimation intend to undergo drug-coated balloon implantation
* Target vessel diameter> 2.5mm

Exclusion Criteria:

* Chronic Total Obstructive lesion
* Diagnose patients with acute myocardial infarction <24 hours
* Can't tolerate or not suitable for RIPC
* Severe hepatic and renal insufficiency
* Expected survival <1 year
* Severe calcification needing rotational atherectomy
* Intolerable to dual antiplatelet therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
TLF | 12 months
  TLF, a composite of cardiac death, target vessel-related myocardial infarction (MI; not clearly attributed to a nontarget vessel and excluding periprocedural MI), or clinically indicated target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Late lumen loss of target vessel（mm） | 6 months
  Late Lumen Loss of target vessel（mm） by Quantitative Coronary Angiography (QCA).
DCB expansion time | less than 120 seconds (On the 1 day of PCI)
  We hypothesis/speculated that the RIPC group had better ischemia tolerance, so the balloon dilation time was longer than the control group.
  But the total time for all patients is less than 120 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai central China cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
After the results are published, researchers can obtain IPD from the responsible person on reasonable request

REFERENCES:
- [Derived] Zhao Z, Yu H, Nie M, Li X, Li M. Remote Ischemic Preconditioning Before Drug-Coated Balloon Implantation can Improve the Long-Term Prognosis of Patients with CAD. Rev Cardiovasc Med. 2024 Mar 27;25(4):116. doi: 10.31083/j.rcm2504116. eCollection 2024 Apr. PMID 39076569